CLINICAL TRIAL: NCT06234358
Title: A Retrospective Observational Clinical Study Carried Out in Patients Operated With Calcanail® in Order to Evaluate the Safety and Performance of the Device
Brief Title: A Clinical Study Carried Out in Patients Operated With Calcanail®
Status: Completed | Type: Observational
Sponsor: FH ORTHO (Industry)
Responsible Party: Sponsor
Other Study IDs: 2017-17
Record Dates: First submitted 2024-01-09; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Calcaneus Fracture; Calcaneus Deformity of Foot; Arthrosis; Localized
MeSH Terms: conditions — Osteoarthritis | interventions — Fracture Fixation, Internal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Calcanail cohort: Patients implanted with medical device under study between January 2012 and January 2020.
  Interventions: Device: osteosynthesis

INTERVENTIONS:
Device: osteosynthesis — calcaneus osteosynthesis is a surgical fixation of a displaced fracture of the calcaneous bone. The surgery is performed under general or regional anesthesia. A scar is made on the lateral side of the ankle below the lateral malleolus. The bone fragments are repositioned as anatomically as possible. They are fixed by a percutaneous nailing fastener.

SUMMARY:
This study is part of the Post-Market Clinical Follow-up process for the Calcanail medical device; the objective of which is to collect data on the safety and performance of the device after it has been placed on the market.

The primary objective of this study is to evaluate the safety of the device. The secondary objectives are to evaluate the clinical performance and safety of the device.

This is a research not involving the human person: observational study, retrospective, monocentric, non-comparative and national.

84 patients will be included in the study.

DETAILED DESCRIPTION:
The CALCANAIL nail is an osteosynthesis nail intended for the repair of articular fractures of the calcaneus, deformities of the hindfoot and arthrosis of the hindfoot. This study aims to answer specific questions about the clinical performance, efficacy or safety of the medical device when used in accordance with its instructions for use. It will also enable us to better detect rare adverse events if necessary, as well as medium-term results.

ELIGIBILITY:
Inclusion Criteria:

1. Patient operated with the studied device between the 01/01/2012 and 01/01/2020.
2. Patient over 18 years old
3. Patient who has received informed information and does not object to the collection of their data in this study.

Exclusion Criteria:

Patient refusing the use of his data or deceased patient who expressed in writing during his lifetime the non-use of his medical information.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient operated with the studied device between the 01/01/2012 and 01/01/2020.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
survival rate (revision) | 12 months
  This objective will be evaluated according to the revision rate in the study

SECONDARY OUTCOMES:
AOFAS score: American Orthopaedic Foot & Ankle Society Score | 12 months
  performance / 100 points represent an "excellent" result and the minimal score was 0
Bone consolidation | 4 months
  Visible on X-ray after surgery
Emergent adverse event | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Julien LUCAS-HERNANDEZ, MD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU Pellegrin, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No